CLINICAL TRIAL: NCT00770757
Title: A Phase 2, Open-Label, Single-Arm, Pilot Study of Safety and Efficacy of CC-4047 (Pomalidomide) in Patients With Advanced Chronic Graft-Versus-Host Disease Developing After Allogeneic Hematological Stem Cell Transplantation
Brief Title: CC-4047 (Pomalidomide) for Graft vs. Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1093 / 201106102
Record Dates: First submitted 2008-10-07; First posted 2008-10-10 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-4047 Arm (Experimental): CC-4047 2 mg orally every day for 1 course (12 weeks or 84 days). Every 28 days of treatment are considered as 1 cycle and every 3 cycles are are considered as 1 course of treatment. A total of 4 courses of treatment are planned (12 months).
  Interventions: Drug: CC-4047

INTERVENTIONS:
Drug: CC-4047
  Other Names: Pomalidomide

SUMMARY:
This study will test the safety and effectiveness CC-4047 (pomalidomide) in patients with advanced, steroid refractory graft-versus-host disease.

DETAILED DESCRIPTION:
Chronic Graft vs. Host Disease is a major complication after allogeneic hematopoietic stem cell transplantation developing in 30 - 70% of patients. It is a multisystem alloimmune and autoimmune disorder with a negative impact on quality of life and functional status, increased need for extended immunosuppression and is the leading cause of late transplant related mortality.

CC-4047 is a novel immune modulatory drug that is a thalidomide analog with a 4,000 fold greater inhibition of TNF-α production related to thalidomide. Several features of CC-4047 suggest that this drug may be useful in treating chronic GVHD including in vitro suppression of TNF-α production, increasing Th1 and stimulation of IL-12 and sIL-Rα.

This study is an open-label, single-arm, pilot study of efficacy and safety of CC-4047 in patients with advanced chronic GvHD who failed to achieve a response with high-dose corticosteroids or second line systemic immunosuppressive therapy.

ELIGIBILITY:
Patient must meet all of the following inclusion criteria:

* Must be greater than or equal to 18 years of age at the time of consent.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Chronic graft versus host disease (GHVD) developing after allogeneic hematological stem cell transplantation diagnosed using NIH criteria for diagnosis and staging of chronic GvHD (including both "classic chronic GvHD" and "overlap syndrome")
* Must have moderate or severe chronic GvHD according to Global Staging System for Chronic GvHD or mild chronic GvHD with platelet count less than 100 x 109/L
* Must have failed to achieve response to high dose corticosteroid (average 0.5 mg/kg/day prednisone or equivalent for greater than or equal to 8 weeks), or have failed second line systemic immunosuppressive therapy.
* If taking corticosteroids at the time of enrollment, must be on stable or tapering schedule without corticosteroid pulses in the preceding 8 weeks.
* If taking secondary systemic immunosuppressive therapy at the time of enrolment, must be on stable or tapering schedule in the preceding 4 weeks.
* Karnofsky performance score (KPS) greater than or equal to 60%.
* Life expectancy greater than or equal to 3 months.
* Female of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse for at least 28 days before starting study drug, while participating in the study, and for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
* FCBP must agree to pregnancy testing and contraceptive counseling every 28 days during the study. FCBP must also refrain from donating blood and/or egg while participating in the study and for at least 28 days after discontinuation from this study
* FCBP must have two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug.
* Must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation.
* Male Subjects must agree to complete abstinence or to use a condom during sexual contact with with a pregnant female or a female of childbearing potential while participating in the study and for at least 90 days following study drug discontinuation even if he has undergone a successful vasectomy
* Must agree to counseling about sexual contact and the potential risks of fetal exposure to pomalidomide every 28 days.
* Male subjects will be warned that sharing study drug is prohibited
* Must agree to abstain from donating blood for at least 28 days following discontinuation of the study drug.
* Must agree to abstain from donating semen or sperm during study participation and for at least 90 days after study drug discontinuation.
* Must agree that if a pregnancy or a positive pregnancy test does occur in a the partner of a male study subject during study participation, the investigator must be notified immediately
* Patients must agree to not share study drug with anyone during participation in the study.
* Must understand and voluntarily sign an informed consent form, or must have a legally authorized representative who is able and willing to voluntarily sign an informed consent form on behalf of the patient.

Exclusion Criteria:

* Pregnant or lactating females.
* New immunosuppressive therapy started within the preceding 4 weeks.
* Extracorporeal photopheresis within the preceding 3 months.
* Hypersensitivity to any immune modulator drug (IMiD™).
* Unable to take prophylactic anticoagulation.
* Any condition which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Acute, persistent, recurrent or late-onset acute GvHD defined by NIH criteria.
* Any of the following laboratory values at registration:

  * absolute neutrophil count (ANC) less than 1.0 x 109/L,
  * platelets less than 75 x 109/L, or
  * creatinine clearance less than 50 mL/min (Cockroft-Gault formula).
* Uncontrolled infection requiring systemic antibiotics.
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection.
* Known uncontrolled arrhythmias or symptomatic heart disease or left ventricular ejection fraction less than 40% (an ECHO should be performed as clinically indicated)
* Recurrence of cancer for which the transplant was done except for presence of minimal residual disease by PCR.
* Other cancer less than or equal to 2 years prior study-entry except:
* Basal cell carcinoma of the skin,
* Squamous cell carcinoma of the skin,
* Carcinoma in situ of the cervix,
* Carcinoma in situ of the breast, or
* Prostate cancer (Tumor, Node, Metastasis [TNM] stage T1a or T1b)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F. DiPersio, M.D., Ph.D., Principal Investigator — Washington Univerisity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/02/2009 and closed to participant enrollment on 03/29/2011.
Period: Overall Study
Arm/Group | CC-4047 Arm
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CC-4047 Arm
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 46 [27 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13
Donor type [Number; unit: participants]
  Matched related donor | 7
  Matched unrelated donor | 6
Karnofsky performance status [Median (Full Range); unit: scores on a scale] — * 90 Able to carry on normal activity; Minor signs or symptoms of disease.
  * 80 Normal activity with efforts; some signs or symptoms of disease.
  * 70 Cares for self; unable to carry on normal activity or to do active work.
  * 60 Requires occasional assistance, but is able to care for most of his personal needs.
  scores on a scale | 80 [60 to 90]
Chronic graft-versus-host disease onset [Number; unit: participants]
  De novo | 5
  Progressive | 1
  Quiescent | 7
Global chronic graft-versus-host disease score [Number; unit: participants] — * Mild - Only 1 or 2 organs or site (except the lung) No clinically significant functional impairment (maximum of score 1 in all affected organs or sites)
  * Moderate - At least 1 organ or site with clinically significant but no major disability (maximum score of 2 in any affected organ or site), or 3 or more organs or sites with no clinically significant functional impairment (maximum score of 1 in all affected organs or sites)
  * Severe - Major disability caused by chronic GvHD (score of 3 in any organ or site) Lung function score ≥ 2
  participants
    Severe | 11
    Moderate | 2
Number of prior therapies [Median (Full Range); unit: number of prior therapies] | 4 [2 to 5]
Years post-transplant [Median (Full Range); unit: years] | 2.5 [1.5 to 15.0]
Years since chronic graft-versus-host disease [Median (Full Range); unit: years] | 1.5 [0.5 to 14.0]
Major organ-systems involved [Number; unit: participants]
  Skin | 13
  Eyes | 10
  Joint and Fascia | 10
  Mouth | 9
  Lungs | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (Complete Response + Partial Response + Other)
Description: * CR is defined as complete resolution in all of signs and symptoms at all affected organs and tissues
  * PR is defined as improvement in greater than or equal to 1 organ/tissue with no progression in any other affected organ/tissue
  * Improvement in chronic GvHD symptoms less than what meets the definition of a PR is defined as other
  * Progressive disease is defined as failure of therapy to control chronic GvHD despite increasing the dose of primary therapy or adding second line treatments
  * No response is defined as no change in disease.
Time Frame: 1 year after last dose of CC-4047
Population: 4 participants discontinued treatment before the third cycle because of adverse-effects and were not evaluable
Measure: Number; unit: participants
Arm/Group | CC-4047 Arm
Number analyzed (Participants) | 9
participants
  Partial overall response | 7
  No response | 2
  Complete overall response | 0
  Progressive disease | 0

2. Secondary Outcome: Safety as Measured by the Most Common Adverse Effects and Reasons for Dose Reductions or Study-discontinuation
Description: -Toxicities will be graded according to the NCI CTCAE v3.0.
Time Frame: 30 days after last dose of CC-4047 or until resolution of event
Measure: Number; unit: participants
Arm/Group | CC-4047 Arm
Number analyzed (Participants) | 13
participants
  Tremors/shakiness | 4
  Muscle cramps/musculoskeletal pain | 12
  Fatigue/anxiety | 6
  Sensory neuropathy | 4
  Respiratory syncytial virus (RSV) pneumonia | 2
  Community-acquired pneumonia | 1
  Sepsis | 1
  Aseptic meningitis | 1
  Deep vein thrombosis/pulmonary embolism | 1
  Erythematous skin rash | 1

3. Post Hoc Outcome: Organ System Response
Time Frame: 1 year after last dose of CC-4047
Population: 4 participants discontinued treatment before the third cycle because of adverse-effects and were not evaluable
Measure: Number; unit: participants
Arm/Group | CC-4047 Arm
Number analyzed (Participants) | 9
participants
  Skin erythema - complete organ response | 2
  Skin erythema - partial organ response | 3
  Skin movable sclerosis - complete organ response | 0
  Skin movable sclerosis - partial organ response | 1
  Mouth - complete organ response | 2
  Mouth - partial organ response | 0
  Eyes - complete organ response | 1
  Eyes - partial organ response | 1
  Gastrointestinal - complete organ response | 2
  Gastrointestinal - partial organ response | 0

4. Post Hoc Outcome: Chronic Graft-versus-host Disease Global Score at the Start/End of the Study
Description: * Global scoring of chronic GvHD consists of questions about various organs including skin, genital tract, lungs, liver, and multiple others. The physician scores each organ from 0 to 3. Score 0 means the patient has no symptoms. Score 1 means the patient has mild symptoms. Score 2 means the patient has moderate symptoms. Score 3 means the patient has severe syptoms.
  * Mild scoring of chronic GvHD is only 1 or 2 organs or site (except the lung). No clinically significant functional impairment (maximum of score 1 in all affected organs or sites)
  * Moderate scoring of chronic GvHD is at least 1 organ or site with clinically significant but no major disability (maximum score of 2 in any affected organ or site) or 3 or more organs or sites with no clinically significant functional impairment (maximum of 1 in all affected orgnas or sites)
  * Severe scoring of chronic GvHD is a major disability caused by chronic GvHD (score of 3 in any organ or site) and lung function score >=2.
Time Frame: 1 year after last dose of CC-4047
Measure: Number; unit: participants
Arm/Group | CC-4047 Arm
Number analyzed (Participants) | 13
participants
  Starting score Severe/Ending score Severe | 11
  Starting score Moderate/Ending score Moderate | 2

5. Post Hoc Outcome: Survival Rate of CC-4047 Responders
Time Frame: Median follow-up 5.6 years (4.2-5.6 years)
Population: Five participants have died and these were the participants who did not respond or were removed from study prior to cycle 3 due to adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | CC-4047 Arm
Number analyzed (Participants) | 7
percentage of participants | 100

ADVERSE EVENTS:
Arm/Group | CC-4047 Arm
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-4047 Arm (N=13)
Abdominal pain (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hypotension (Vascular disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
RSV infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (General disorders) | 1
Tremors (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-4047 Arm (N=13)
Albumin - low (Metabolism and nutrition disorders) | 7
Alkaline phosphatase (Investigations) | 6
Allergic reaction/hypersensitivity (Immune system disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Anal incontinence (intermittent) (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blistering/tenderness/erythema/desquamating rash (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Calcium - low (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine (Renal and urinary disorders) | 2
Decreased range of motion (joint function) (Musculoskeletal and connective tissue disorders) | 3
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Distension/bloating (Gastrointestinal disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Edema (General disorders) | 1
Edema (generalized) (General disorders) | 1
Edema (limb) (General disorders) | 2
Fatigue (General disorders) | 4
Fracture (Injury, poisoning and procedural complications) | 1
Fracture of vertebra (compression) (Injury, poisoning and procedural complications) | 1
Glucose - high (Metabolism and nutrition disorders) | 8
Glucose - low (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 9
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection without neutropenia (Infections and infestations) | 6
Lymphopenia (Investigations) | 9
Magnesium - high (Metabolism and nutrition disorders) | 1
Magnesium - low (Metabolism and nutrition disorders) | 2
Mood alteration - anxiety (Psychiatric disorders) | 3
Mood alteration - depression (Psychiatric disorders) | 1
Mucositis - mouth sensitivity (Gastrointestinal disorders) | 1
Mucositis - oral ulcers (Gastrointestinal disorders) | 3
Muscle pain (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 1
Nephrolithiasis - passing stones (Renal and urinary disorders) | 1
Neuropathy - sensory (pain) (Nervous system disorders) | 1
Neuropathy - motor (weakness) (Nervous system disorders) | 1
Neuropathy - sensory (numbness) (Nervous system disorders) | 2
Neutrophils (ANC) (Investigations) | 1
Osteonecrosis (avascular) (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain NOS (General disorders) | 1
Platelets (Investigations) | 2
Potassium - low (Metabolism and nutrition disorders) | 4
RSV infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
SGOT (AST) (Investigations) | 9
SGPT (ALT) (Investigations) | 11
Sclerodermatous fibrosis (Skin and subcutaneous tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Skin wound/break (Skin and subcutaneous tissue disorders) | 1
Sodium - high (Metabolism and nutrition disorders) | 3
Sodium - low (Metabolism and nutrition disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/embolism (Vascular disorders) | 1
Tremor (Nervous system disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Wrist pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes